CLINICAL TRIAL: NCT06141499
Title: Using Shared Decision Making to Improve Kidney Transplantation Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Kidney Transplant Collaborative (Unknown); National Kidney Foundation, United States (Other)
Responsible Party: Principal Investigator, Sumit Mohan, MD, Professor of Medicine and Epidemiology, Columbia University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAU1202
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: End Stage Renal Disease; Kidney Failure
Keywords: Kidney Transplant; Transplantation; Shared Decision Making
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: Enrolled providers and enrolled patients will receive different interventions; outcomes assessed for these two groups will be different.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Providers (Experimental): Dialysis providers will receive educational material about the kidney transplantation and waitlisting process.
  Interventions: Behavioral: Provider educational materials
- Patients (Experimental): Dialysis patients will receive letters with information about their status within the kidney transplantation and waitlisting process.
  Interventions: Behavioral: Patient letters

INTERVENTIONS:
Behavioral: Provider educational materials — Dialysis providers will receive educational material about the kidney transplantation and waitlisting process.
  Arms: Providers
Behavioral: Patient letters — Dialysis patients will receive letters with information about their status within the kidney transplantation and waitlisting process. Letters will describe kidney waitlist status, living donor transplantation, Hepatitis C positive kidney transplants, and high Kidney Donor Profile Index (KDPI) transplants.
  Arms: Patients

SUMMARY:
The goal of this clinical trial is to increase shared decision-making between dialysis providers and patients in order to increase patients' probability of transplantation and to reduce socioeconomic/racial disparities in access to kidney transplantation.

Participants will receive educational material over the course of 4-6 months about different aspects of the kidney transplant and waitlisting process.

DETAILED DESCRIPTION:
Kidney transplantation is the preferred treatment choice for patients with end stage kidney disease (ESKD), yet only a small proportion of patients with incident ESKD are counseled about their transplant options. Often, a smaller minority of patients reach the transplant waitlist in a timely manner. Increasing the likelihood of transplantation for patients with ESKD can lead to longer survival, better quality of life, and reduced costs of care.

The kidney transplant and waitlist process is a complex and multi-step process that occurs over an extended period of time. This process involves transitions of care between multiple providers and requires patients to be proactive in their medical evaluations.

This study will deliver educational materials to dialysis care teams and provide quarterly, personalized informational letters to patients, with the aim of increasing shared decision-making between patients and providers by giving them the information needed to initiate conversations about kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* On a waitlist or undergoing an evaluation at the Columbia University/New York Presbyterian Hospital (CU/NYPH) Transplant Center or at the Cleveland Clinic (CC)
* Receiving hemodialysis at one of the following dialysis clinics:

  * Fresenius Kidney Care City Dialysis
  * DaVita Kidney Care Haven Dialysis
  * DaVita Melrose Dialysis
  * DaVita Highbridge Dialysis
  * Rogosin Institute East Side Dialysis Unit
  * Rogosin Institute West Side Dialysis Unit

Exclusion Criteria:

* Speaking a language other than English or Spanish
* Younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Change in patient knowledge of individual waitlist status | Baseline (day 1), post letter 1 (approx 1 month later), post letter 2 (approx 1 month later), post letter 3 (approx 1 month later), post intervention (approx 4-6 months total)
  Patient knowledge of individual waitlist status will be measured by one Yes/No question on the patient survey using McNemar's test.
Change in frequency of shared decision-making conversations, | Baseline (day 1), post letter 1 (approx 1 month later), post letter 2 (approx 1 month later), post letter 3 ( approx 1 month later), post intervention (approx 4-6 mos total)
  Frequency of shared decision-making conversations will be measured by two Yes/No questions on the patient survey using McNemar's test.
Change in donor kidney preferences | Baseline (day 1), post letter 1 (approx 1 month later), post letter 2 (approx 1 month later), post letter 3 (approx 1 month later), post intervention (approximately 4-6 mos total)
  Patient preferences for kidneys from living donors, kidneys from Hepatitis C positive donors, and kidneys from high KDPI donors will be measured by six Yes/No questions on the patient survey using McNemar's test.

SECONDARY OUTCOMES:
Change in dialysis provider attitudes, as measured on provider survey | Post-educational session, Day 1
  Dialysis providers' attitudes and comfort with discussing the kidney waitlist and transplantation process will be measured on the provider survey. Questions will be scored on a 1-5 Likert scale, with 1 indicating low comfort level and 5 indicating high comfort level. Total scores range from 5-25 with a higher score indicating a better outcome.
Provider assessment of patient letters, as measured on provider survey | End of intervention/at completion of letter delivery (4-6 months)
  Providers' assessment of the helpfulness of patient letters will be measured by five questions on the provider survey. Questions will be scored on a 1-5 Likert scale, with 1 indicating low helpfulness and 5 indicating high helpfulness. Total scores range from 5-25 with a higher score indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sumit Mohan, MD, MPH, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University, New York, New York
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No